CLINICAL TRIAL: NCT04180813
Title: A Non-interventional Study of Patient Medication Adherence and Treatment Effectiveness Among New Users of Linagliptin and Acarbose in the Real-world Clinical Setting in China
Brief Title: Real-world Study Comparing the Adherence and Effectiveness of Linagliptin vs. Acarbose
Status: Terminated | Type: Observational
Why Stopped: Study enrollment did not meet expectation.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1218-0184
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; Acarbose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Linagliptin Initiators
  Interventions: Drug: Linagliptin
- Acarbose Initiators
  Interventions: Drug: Acarbose

INTERVENTIONS:
Drug: Linagliptin — drug
  Other Names: Trajenta®
  Groups: Linagliptin Initiators
Drug: Acarbose — drug
  Groups: Acarbose Initiators

SUMMARY:
Non-interventional cohort study based on newly collected data under routine medical practice of a total of 500 Diabetes Mellitus, Type 2 patients

ELIGIBILITY:
Inclusion Criteria:

* Patient should fully know and understand the content of consent form, and the patient is willing and able to sign an informed consent form
* Chinese outpatients with confirmed T2DM
* Patients of ≥ 18, < 80 years old
* Patients currently use metformin monotherapy ≥ 1500 mg/day or maximum tolerable dose and whose glucose levels are not adequately controlled
* HbA1c ≥ 7% and < 12%
* New user* linagliptin or acarbose as combination therapy with metformin ≥ 1500 mg/day or maximum tolerable dose *New user defined as a T2DM patient initiating linagliptin or acarbose as an add-on therapy.

These are patients who are on metformin and whose glucose levels are not adequately controlled.

Exclusion Criteria:

* Type 2 diabetes mellitus patients who previously used any DPP-4 inhibitor/ GLP-1 receptor agonist at index date or any AGI at index date, are not eligible to participate. Also excluded are patients who currently using any glucose-lowering agent as monotherapy other than metformin.
* Patients with clinically significant acute major organ or systemic disease or other condition judged by the investigator that would create difficulty for the 24-week follow-up.
* Patients who participated in a clinical trial within 2 months prior to study enrolment date.
* Patients diagnosed with Type 1 diabetes mellitus, secondary diabetes or gestational diabetes.
* Current treatment with systemic steroids at time of informed consent or within 6 weeks prior to informed consent.
* Patients with known significant GI disease as judged by the study physician.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 500 outpatients with T2DM from 16 sites distributed in different regions in mainland China.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2021-07-11 (Actual); Study Completion 2021-07-11 (Actual)

PRIMARY OUTCOMES:
Proportion of T2DM patients with high medication adherence at Week 24 | 24 weeks

SECONDARY OUTCOMES:
The effectiveness of linagliptin and acarbose on glycemic control evaluated by reducing HbA1c during a 24 week follow-up in two groups | 24 weeks
Proportion of T2DM patients achieving a therapeutic glycemic response defined as HbA1c < 7.0% or a lowering of HbA1c ≥ 0.5% | 24 weeks
To compare the composite endpoint (proportion of achieving HbA1c < 7.0% without gastrointestinal adverse events (GI AEs) and without an investigator defined hypoglycaemic event) | 24 weeks
Patient satisfaction by Diabetes Treatment Satisfaction Questionnaire (DTSQ) among linagliptin and acarbose initiators. The DTSQ would be completed at routine physician visits since initiation of the drug | 24 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - No.731 Hospital of China Aerospace Science & Industry Corp., Beijing
  - Affiliated Hospital of Chengdu University, Chengdu
  - ChongQing The Fourth Hospital, Chongqing
  - Dongying People's Hospital, Dongying
  - Huai'an first people's hospital, Huai'an
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - Shanghai TCM-Integrated Hospital, Shanghai
  - Southern Medical University Shenzhen Hospital, Shenzhen
  - Zhangjiagang First People Hospital, Suzhou

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com